CLINICAL TRIAL: NCT03635307
Title: Ability of Changes in End Tidal Carbon Dioxide to Assess the Stroke Volume Effects of a Volume Expansion of 250ml of Crystalloid in the Operating Room
Acronym: REVCO2
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/18
Record Dates: First submitted 2018-08-08; First posted 2018-08-17 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Blood Volume Expansion
Keywords: Blood Volume expansion; Fluid responsiveness; Stroke volume; Perioperative optimization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Operated patients with volume expansion
  Interventions: Other: End Tidal Carbon Dioxide measure

INTERVENTIONS:
Other: End Tidal Carbon Dioxide measure — End Tidal Carbon Dioxide measures before and after a volume expansion of 250ml of crystalloid in the operating room.

SUMMARY:
Volume expansion is the cornerstone of perioperative hemodynamic optimization. The main objective of volume expansion is to increase and to maximize stroke volume. Despite national and international recommendations, stroke volume monitoring is clearly not widely adopted. This is mostly due to the cost and the invasiveness of the devices allowing stroke volume monitoring. End tidal carbon dioxide is monitored in all patients undergoing general anaesthesia and is totally non-invasive. A strong relationship between stroke volume and end tidal carbon dioxide have been already demonstrated. The aim of the present study is to determine if change in End Tidal Carbon Dioxide can assess the stroke volume effects of a volume expansion of 250ml of crystalloid in the operating room

DETAILED DESCRIPTION:
The main objective of volume expansion is to increase stroke volume. Franck-Starling curve is schematically divided into two portions: a vertical portion which mean that an increase in preload secondary to volume expansion will induce an increase in stroke volume; and a flat portion which mean that a same increase in preload will not induce an increase in stroke volume. Perioperative optimization is based on stroke volume maximization using volume expansion. Despite national and international recommendations, stroke volume monitoring is clearly not widely adopted. This is mostly due to the cost and the invasiveness of the devices allowing stroke volume monitoring. End tidal carbon dioxide is monitored in all patients undergoing general anaesthesia and is totally non-invasive. Several studies evaluated the relationship between stroke volume and end tidal carbon dioxide and other studies evaluated the ability of changes in end tidal carbon dioxide to assess changes in stroke volume induced by volume expansion with discordant results. These studies included small sample size and were heterogeneous (intensive care unit and nor operating room, volume expansion or passive leg raising, crystalloid or colloid, 500ml and not 250 ml ….). Nowadays, it is not clear if changes in end tidal carbon dioxide can be considered as a surrogate of changes in stroke volume during a volume expansion in operating room patients. Thus, the aim of the present study is to determine if change in End Tidal Carbon Dioxide can assess the stroke volume effects of a volume expansion of 250ml of crystalloid in the operating room.

The follow up will be restricted to the duration of volume expansion. The last data will be collected just after the end of volume expansion.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years
* Scheduled for neurosurgery in prone position
* Equipped from an arterial catheter and stroke volume monitoring

Exclusion Criteria:

Patient with cardiac dysfunction and/or lung disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient older than 18 years scheduled for neurosurgery in prone position, equipped from an arterial catheter and stroke volume monitoring in Bordeaux University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
End Tidal Carbon Dioxide measure | Beggining time of volume expansion of 250ml of crystalloid during surgery
End Tidal Carbon Dioxide measure | 1 minute after the end of volume expansion of 250ml of crystalloid during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Courson H, Chauvet J, Le Gall L, Georges D, Boyer P, Verchere E, Nouette-Gaulain K, Biais M. Utility of changes in end-tidal carbon dioxide after volume expansion to assess fluid responsiveness in the operating room: a prospective observational study. Br J Anaesth. 2020 Nov;125(5):672-679. doi: 10.1016/j.bja.2020.07.018. Epub 2020 Aug 27. PMID 32863016